CLINICAL TRIAL: NCT05905211
Title: Investigation of the Balance, Functional Mobility, Quality of Life, Fear of COVID-19 and Emotional State of the Elderly Infected and Non-Infected With COVID-19
Brief Title: Investigation of Physical and Emotional Status the Elderly Infected and Non-Infected With COVID-19
Status: Completed | Type: Observational
Sponsor: Tarsus University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ali MUTLU, Research Assistant, Tarsus University
Other Study IDs: TU-FTR-AMUTLU-1
Record Dates: First submitted 2023-06-12; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Pandemic
Keywords: Geriatrics; Aged; Functional Status; Postural Balance; Quality of Life; Activities of Daily Living; Fear; Depression; COVID-19
MeSH Terms: conditions — COVID-19; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected COVID-19: Balance, functional mobility, activities of daily living, quality of life, fear of COVID-19, depression evaluated
  Interventions: Other: Observational Tests
- Non-Infected COVID-19: Balance, functional mobility, activities of daily living, quality of life, fear of COVID-19, depression evaluated
  Interventions: Other: Observational Tests

INTERVENTIONS:
Other: Observational Tests — The Berg Balance Scale was used to evaluate the balance levels, the Timed Up and Go Test was used to evaluate the functional mobility levels, and the Functional Independence Scale was used to evaluate the activities of daily living. The World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD) was used to evaluate the quality of life, the Fear of COVID-19 Scale was used to evaluate the COVID-19 fear levels, the Geriatric Depression Scale was used to evaluate the symptoms of depression.

SUMMARY:
The aim of this observational study is to evaluate individuals in terms of balance, functional mobility, influences in activities of daily living, fear of COVID-19, moods, quality of life parameters in order to investigate the effects of COVID-19 on elderly individuals.

DETAILED DESCRIPTION:
This study was carried out to investigate the status of elderly individuals who survived the COVID-19 in terms of different parameters such as balance, functional mobility, activities of daily living, quality of life, fear of COVID-19, depression. A total of 107 elderly individuals aged 65 and over were included in the study, including 52 elderly individuals who survived the COVID-19 and 55 elderly individuals who non-infected COVID-19. The sociodemographic information of the participants was recorded. The Berg Balance Scale was used to evaluate the balance levels, the Timed Up and Go Test was used to evaluate the functional mobility levels, and the Functional Independence Scale was used to evaluate the activities of daily living. The World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD) was used to evaluate the quality of life, the Fear of COVID-19 Scale was used to evaluate the COVID-19 Fear levels, the Geriatric Depression Scale was used to evaluate the symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Being an individual aged 65 and over voluntarily to participate in the study
* Not having a problem affecting understanding and speaking, having the ability to walk without any help

Exclusion Criteria:

* Having any musculoskeletal or neurological problem that may affect walking and balance
* Have a known mental problem

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Including 52 elderly individuals who survived the COVID-19 and 55 elderly individuals who non-infected COVID-19.
  The group who had COVID-19 was treated in the pandemic ward of Tarsus State Hospital with a definitive diagnosis of COVID-19, and over whose condition was planned to be discharged were included in the study just before discharge.
  Elderly individuals aged 65 and over who did not have COVID-19 were reached in Tarsus city center by snowball sampling method.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 2 months
  It is a method that allows functional assessment of balance in individuals through activities of daily living. Its Turkish validity and reliability was conducted by Sahin et al. The scale consists of 14 items that the researcher fills in by observing the individual and each item is graded between 0 and 4 points. It includes daily functional activities such as standing up from a sitting position, standing and sitting without support, reaching forward while standing, picking up objects from the floor, turning 360°, standing on one leg. A ruler, stopwatch, chair, step, etc. are used during the test. The highest score that can be obtained from the test is 56 and the range of 0-20 points indicates a balance disorder leading to a high risk of falling, the range of 21-40 points indicates that the individual has an acceptable balance, and the range of 41-56 points indicates that the individual has good balance.
Timed Up and Go Test | 2 months
  It is a reliable method widely used to assess functional mobility and balance in individuals. It is a test that the researcher applies by observing the individual. The test starts with the command "start" and ends with the participant getting up from the chair, walking 3 meters, turning around and then walking back to the chair and sitting down. The time from the "start" command to the end of the test is measured with a stopwatch.
Functional Independence Scale | 2 months
  It shows the independence levels of individuals in basic physical and cognitive functions in activities of daily living. Turkish validity and reliability was conducted by Kücükdeveci et al. The scale is administered by the researcher's observation of the physical condition and question and answer method. It measures two sub-headings: physical/motor function and cognitive/cognitive function. In the scale consisting of 18 items in total, 13 questions evaluate motor functions and 5 questions evaluate cognitive functions. Self-care, sphincter control, transfer, mobility, communication, social perception are the functions questioned by the scale. Each item is scored between 1-7 points. 7 points indicates complete independence and 1 point indicates complete dependence. The participant can score between 18-126 points on the scale. A high total score indicates a high level of independence.
The World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD) | 2 months
  It is a six-dimensional, 5-point Likert-type scale consisting of 24 questions and used to assess quality of life in the elderly. Its Turkish validity and reliability was performed by Eser et al. (2010) The scale is applied in the form of question and answer. The sub-dimensions of the scale are sensory functions, autonomy, past-present and future activities, social participation, dying and death, and closeness. Scoring for each question is done on a scale of 1-5. Possible dimension scores range from 4-20. In addition, a total score can be calculated by adding the scores together. A higher score indicates an improved quality of life.
The Fear of COVID-19 Scale | 2 months
  It is a unidimensional scale and consists of a total of 7 items, each item is designed in 5-point Likert type. The scale was adapted into Turkish by Bakioglu et al. (2021). The scale is applied in question and answer form. The participant is asked to mark between '1 - Strongly Disagree' and '5 - Strongly Agree'. A score between 7-35 is obtained from the scale. An increase in the total score indicates that the participant's level of fear of COVID-19 has increased.
Geriatric Depression Scale | 2 months
  It is a self-report scale consisting of a total of 30 questions that should be answered yes/no. Its Turkish validity and reliability was conducted by Ertan et al. (1997). The minimum score that can be obtained in the scale is 0 and the maximum score is 30, and each answer given for depression status is 1 point and the other answers are 0 points. A score range of 0-10 points indicates no depression, a score range of 11-13 points indicates possible depression, while scores of 14 points and above are considered as definite depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ali MUTLU, Principal Investigator — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No